CLINICAL TRIAL: NCT00911352
Title: Nurse-initiated Cryotherapy Intervention for Docetaxel-induced Nail Toxicities: Case-control Study
Brief Title: Cryotherapy Intervention for Docetaxel-induced Nail Toxicities
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Princess Alexandra Hospital, Brisbane, Australia (Other)
Responsible Party: Principal Investigator, Alexandra McCarthy, Associate Professor, Princess Alexandra Hospital, Brisbane, Australia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009/043
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Effects of Chemotherapy
Keywords: Cryotherapy; Hand toxicity; Nail toxicity; Infection control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Frozen gel glove (Elasto-Gel Mitten) (Experimental): Cryotherapy hand
  Interventions: Device: Frozen gel glove (Elasto-Gel Mitten)
- No frozen glove therapy (No Intervention): Usual care

INTERVENTIONS:
Device: Frozen gel glove (Elasto-Gel Mitten) — Gel glove is frozen for > 3 hours at -5 to -30°C prior to use. Each patient wears a triple glove set (surgical glove overlaid with cotton glove, overlaid with gel glove) on their intervention hand. Gloves are worn for duration of infusion (15 mins pre, 60 minutes intratreatment and 15 mins post) to ensure the patients' peripheries are vasoconstricted on commencement of the infusion and for enough time afterwards to ensure circulating drug does not reach the target area. Because of the duration of the infusion, more than one gel glove will be used successively (for 45 minutes each) to maintain a consistently low temperature on the hand and nails.
  Other Names: Elasto-Gel Mitten
  Arms: Frozen gel glove (Elasto-Gel Mitten)

SUMMARY:
Between 30% and 88% of chemotherapy patients receiving docetaxel experience side effects of the hand ranging from skin and nail disfigurement, blistering, desquamation, pain, infection, and impaired treatment-related quality of life and function. Preliminary data indicate that nurse-initiated cryotherapy during treatment may lower the incidence and severity of these side effects, but several issues should be addressed before this intervention is implemented in hospital settings. These include more rigorous study design, larger sampling frames, and consideration of infection control concerns. This study will address these issues, thereby rigorously evaluating the safety and efficacy of nurse-initiated cryotherapy at Princess Alexandra Hospital.

DETAILED DESCRIPTION:
Research problem:

Internationally, cryotherapy for docetaxel-induced nail and skin toxicities of the hand has become a popular primary treatment. Yet there is little evidence beyond one Phase II, non-randomised, (n=45) study to support such widespread use. There are also unanswered concerns relating to the potential of this treatment to cross-infect patients at risk of immunocompromise. This phase II case-control study extends previous work to address sample size concerns, enhance methodological rigour and add new evidence with respect to infection control, prior to its possible implementation at Princess Alexandra Hospital (PAH).

Hypothesis/questions/outcomes:

Aim: This study will investigate the utility, efficacy and safety of cryotherapy, in the form of frozen gel gloves, with respect to the prevention of docetaxel-induced nail and skin toxicities in cancer patients.

Hypotheses:

H1: Cryotherapy reduces the incidence and severity of docetaxel-induced nail and skin toxicities.

H2: Cryotherapy to prevent docetaxel-induced nail and skin toxicities is tolerated by cancer patients.

H3: A standardised decontamination protocol prevents healthcare-acquired infections potentially associated with cryotherapy.

Anticipated results: The primary endpoint is a decrease in the incidence and severity of nail and skin toxicities over the course of treatment, as measured by the CTCAE scores. Secondary endpoints include delayed time to occurrence of any nail or skin toxicity; patient comfort; and a successful glove decontamination protocol as evidenced by the absence of epidemiologically significant organisms on frozen gloves.

Research design:

Population and sampling: Approximately 300 new breast, prostate and lung cancer patients are diagnosed per year at PAH. Not all of these are treated with docetaxel, and some are placed on clinical trials, so will not be available for enrolment in the study. Data from PAH Human Information Management Services indicates that approximately 120 patients will therefore be eligible to enrol in the study. Accounting for a 50% rate of refusal or failure to meet the study criteria, it is anticipated that approximately 60 patients will enrol in the study in 12 months. This amounts to 60 control and 60 intervention hands for comparison.

Withdrawal criteria: severe cold intolerance or withdrawal of consent.

Procedure: Standard cryotherapy comprises a disposable cotton glove overlaid with a glycerine gel-filled glove, which cover the hand to the wrist and separate the thumb from the rest of the hand. The gel glove is frozen for at least 3 hours at -0.25 to -0.30°C prior to use. Each patient's hands will be randomly allocated to intervention or control. Each patient will wear the triple glove set on their intervention hand. No glove set will be used on the other hand, which acts as the case control. During each docetaxel infusion, the patient will wear the gloves for a total of 90 minutes (15 minutes before the administration of docetaxel, during the 1-hour docetaxel infusion, and 15 minutes after the end of infusion). This is a standard procedure during cryotherapy that will ensure the patients' peripheries are vasoconstricted on commencement of the infusion and for enough time afterwards to ensure circulating drug does not reach the target area. Because of the duration of the infusion, more than one gel glove will be used successively (for 45 minutes each) to maintain a consistently low temperature on the hand and nails. Using this method, the study will determine the comparative incidence of skin and nail disorders with and without cold protection.

The additional infection control measure in this study incorporates (1) insertion of a disposable surgical glove (which exceeds the length of the cotton and gel gloves) between the cotton and gel gloves to minimise the risk of cross-contamination and (2) surface decontamination using a standard cleaning protocol. The term 'cleaning' refers to the use of mechanical action, detergent and warm water, followed by rinsing and drying. It aims to remove organic matter, visible soils and salts from the glove surface. Cleaning removes the bulk of micro-organisms from surfaces and they are also unable to multiply on inanimate surfaces cleaned and dried in this manner. In accordance with the Spaulding Classification System the glove cleaning protocol will incorporate 1) cleaning all internal and external surfaces with neutral detergent and warm water; 2) rinsing with clean water; 3) cleaning all internal and external surfaces with a 70% alcohol-based solution; and 4) complete air drying of the glove.

Data collection: Patients receive docetaxel once every 21 days for 126 - 189 days (i.e. on 6 to 9 separate occasions each; docetaxel is administered on day 1 of each cycle). Nail and skin toxicity appear between days 36 to 72 in untreated patients, and increases in severity until the end of treatment2-6,8. Cryotherapy will commence on day 1; will occur every 21 days with docetaxel administration thereafter, and cease after the final dose of docetaxel. Patients' toxicities will be assessed independently prior to the commencement of each of the docetaxel infusions, and three-weekly thereafter, by 2 blinded clinical nurse assessors using the Common Toxicity Criteria for Adverse Events1. The assessors will be trained by a dermatologist in the rating of these toxicities prior to study commencement. The training will also establish inter-rater reliability ratings between assessors, using digital photographs of skin and nail toxicities already available from clinical trials records at Princess Alexandra Hospital. In addition to blinded in-clinic assessment, digital photography of each hand will be undertaken under standardised lighting conditions prior to the commencement of each infusion. This will enable the nurses' assessment to be regularly compared with the dermatologist's assessment to ensure inter-rater reliability.

Because the final infusion may also affect the nails beyond treatment cessation, nail assessment will also be undertaken 3 weeks after the last infusion during routine OPD follow-up. Patients' comfort level with cryotherapy will also be assessed during each of the infusions, using a 4-point rating system to determine whether patients are dissatisfied (0), not very satisfied (1), satisfied (2), or very satisfied (3) with the treatment in terms of glove contact, temperature tolerance and immobilisation constraints.

A pre-post assessment of the decontamination protocol of the gel glove at each of the treatment sessions will also be undertaken. Microbial Cultural and Sensitivity (MC&S) and antibiograms will be undertaken on swabs taken from glove surfaces at T1 (pre-decontamination) and T2 (post- decontamination). Sites for swabbing of all gloves will be standardised to 1) the internal glove surface of the back of the hand; 2) the internal glove surface of the palm of the hand; 3) the internal glove surface at the tip of the second index finger; and 4) the internal glove surface at tip of the thumb. These sites are well-established as being problematic for cleaning and decontamination in hand hygiene, where carriage of microbial organisms is high31. MC&S and antibiograms will test for non-multidrug-resistant Staphylococcus Aureus (nmMRSA); multidrug-resistant Staphylococcus Aureus (MRSA), and vancomycin-resistant Enterococcus, extended spectrum (VRE).

A client record form will record and update relevant demographic, disease- and treatment-related data at each time point.

Data analysis:

Analyses of skin and nail toxicity will replicate the method used in the original study, and will be undertaken on an intention-to-treat basis. Matched-pair t-tests will be used to determine the statistical significance of any differences in the incidence and severity of nail and skin toxicities between protected and unprotected hands. Because time-to-event endpoints will be used, Kaplan-Meier and log-rank methods will estimate differences in time to toxicity occurrence. The impact of nail and skin toxicity occurrence for confounders and covariates will be determined via multivariate Cox regression analyses. Frozen glove contamination will be analysed by determining frequencies and types of micro-organisms.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving docetaxel as mono- or combination therapy
* patients with no nail disorders at the start of treatment
* life expectancy of at least 3 months

Exclusion Criteria:

* patients previously treated with taxane chemotherapy
* Raynaud's phenomenon
* distal metastases
* ungual pathology
* arteriopathy
* cold intolerance
* peripheral neuropathy of grade 2 or higher
* patients currently enrolled in clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Differences in the incidence and severity of nail and skin toxicities between protected and unprotected hands | 12 months

SECONDARY OUTCOMES:
Safety and tolerability of frozen glove treatment | 12 months
Adequacy of infection control measure added to glove protocol | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra McCarthy, PhD, Principal Investigator — Queensland University of Technology
Locations (1):
- Princess Alexandra Hospital, Woolloongabba, Queensland, Australia

REFERENCES:
- [Derived] McCarthy AL, Shaban RZ, Gillespie K, Vick J. Cryotherapy for docetaxel-induced hand and nail toxicity: randomised control trial. Support Care Cancer. 2014 May;22(5):1375-83. doi: 10.1007/s00520-013-2095-x. Epub 2013 Dec 22. PMID 24362908